CLINICAL TRIAL: NCT04608669
Title: Transient Acetaminophen Induced Hypothermia in Pediatrics Population Undergoing General Anesthesia
Brief Title: Paracetamol Hypothermia Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saint George Hospital (Other)
Responsible Party: Principal Investigator, Hazem Kafrouni, Assistant professor, Saint George Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SaintgeorgeHh
Record Dates: First submitted 2020-10-24; First posted 2020-10-29 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Safety Issues
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temperature comparison (Other)
  Interventions: Drug: Paracetamol
- No change (Active Comparator)
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol — Give paracetamol or placebo and compare temperature

SUMMARY:
Transient Acetaminophen Induced Hypothermia in Pediatrics Population Undergoing General Anesthesia

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Ages: 0 Days to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Temperature variation | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Georges hospital, Beirut, Lebanon